CLINICAL TRIAL: NCT00638495
Title: Phase II Study of TRK-820 Soft Capsules - Intractable Pruritus in Patients With Chronic Liver Disease -
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Toray Industries, Inc, Pharmaceutical Clinical Research Dept.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 820HPC01
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2010-01

CONDITIONS: Pruritus With Chronic Liver Disease
MeSH Terms: interventions — TRK 820

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Nalfurafine Hydrochloride (TRK-820)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nalfurafine Hydrochloride (TRK-820) — TRK-820 2.5, 5 and 10 microg is to be administered orally once daily, after supper in principle, for 28 days.
  Other Names: REMITCH
  Arms: 1
Drug: Placebo — Placebo is to be administered orally once daily, after supper in principle, for 28 days.
  Arms: 2

SUMMARY:
The efficacy and safety of TRK-820 are to be evaluated in the treatment of intractable pruritus in patients with Chronic Liver Disease by administering 2.5, 5 and 10 microg of this drug or placebo for 28 days in four groups with a design of randomized, double-blind, parallel-group comparison. In addition, the plasma concentrations of TRK-820 and its primary metabolites are to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Liver Disease is present; and the patient's general condition is judged by the physician to be stable with no prospect of an abrupt change in pathophysiology.
* It can be confirmed by either of the following that treatment of pruritus with antihistamines or antiallergics has not been adequately effective in such patients:

Exclusion Criteria:

* Malignant tumors
* Depression, integration dysfunction syndrome (schizophrenia), or dementia
* Hepatic encephalopathy, or hepatic cirrhosis in which ascites or esophageal or gastric aneurysm cannot be controlled
* Alcoholic liver disease
* Atopic dermatitis, chronic urticaria, or other skin disease producing generalized pruritus that is judged by the physician to affect the assessment of pruritus associated with Chronic Liver Disease in this study
* Allergy to opioid drugs
* Drug dependence or alcohol dependence
* Chronic renal failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in VAS value (based on morning or evening scores, whichever larger, during the treatment period [4th week]) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Toray Industries, Inc, Urayasu, Chiba, Japan